CLINICAL TRIAL: NCT06182878
Title: A Single-arm Trial of a Web Based TLC (Tender Loving Care) Platform to Psychologically Support Patients With Recurrent Pregnancy Loss
Brief Title: Tender Loving Care for Recurrent Pregnancy Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-17302
Record Dates: First submitted 2023-11-28; First posted 2023-12-27 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Recurrent Pregnancy Loss
Keywords: Recurrent Pregnancy Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tender loving care intervention (Experimental): Weekly prenatal counseling messages sent via an online platform.
  Interventions: Behavioral: Tender loving care intervention

INTERVENTIONS:
Behavioral: Tender loving care intervention — Receiving weekly prenatal care counseling messages

SUMMARY:
The goal of this investigational study is to evaluate participation in a weekly, interactive, tender loving care messaging platform impact on pregnancy outcomes in patients with recurrent pregnancy loss.

The main questions it aims to answer are: (1) does participation in weekly, interactive tender loving care messages increase live birth rates in patients with recurrent pregnancy loss? (2) Does participation in weekly, interactive tender loving care messages increase patients' quality of life? Does participation in weekly, interactive tender loving care messages decrease patients' depressive symptoms?

Participants will be asked to interact with weekly messages providing prenatal counseling and support. Additionally, patients will be asked to complete the fertility quality of life survey several times over the course of the pregnancy.

DETAILED DESCRIPTION:
Participants will be asked to interact with weekly messages providing prenatal counseling and support. Additionally, patients will be asked to complete the fertility quality of life survey several times over the course of the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals receiving their prenatal care at WRNMMC
* Able to speak and understand English
* Less than or equal to 10+0 weeks gestation by last menstrual period (LMP) or dating ultrasound at the time of enrollment
* At least two prior pregnancy losses. Pregnancy losses must be confirmed with laboratory criteria confirming a positive pregnancy test in the military electronic medical record with subsequent resolution (resolution may be reported by patient), or with ultrasound criteria demonstrating an intrauterine gestational sac with subsequent resolution (resolution may be reported by patient).

Exclusion Criteria:

* Age less than 18 years and older than 44 at time of enrollment
* Unable to speak or understand English
* Current smoker or tobacco use within 30 days
* History of uterine anomaly, coagulopathy, balanced translocation, endometrial polyps, submucosal fibroids, pathology confirmed acute or chronic endometritis, hydrosalpinx, history of Asherman syndrome, poorly controlled endocrinopathies, HIV infection
* History of gonadotoxic therapy or cancerous condition of the female reproductive tract
* Suspicion for or confirmation of an ectopic pregnancy

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Live birth rates | through study completion, an average of 1 year
  Live birth is defined as the delivery of at least one live-born infant at or after 22+0 weeks gestational age

SECONDARY OUTCOMES:
Fertility quality of life survey scores | Baseline at enrollment of study, repeat assessments at 13 weeks, 28 weeks, and 6 weeks after delivery or after miscarriage
  Quality of life will be defined using the fertility quality of life scores. The survey is entitled, "Fertility quality of life questionnaire." Survey responses are based on a five-point scale, with responses such as "very good" and "very satisfied" corresponding to better outcomes.
Depressive symptoms | through study completion, an average of 1 year
  Depressive symptoms will be defined using the survey entitled, "Edinburgh Postnatal Depression Scores." This survey uses a four-point scale for each response, with higher cumulative scores corresponding to worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: David Boedeker, DO, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No